CLINICAL TRIAL: NCT06578104
Title: PULSED AF Post-Approval Study, an Addendum to the PulseSelect™ PFA Global Registry
Brief Title: PULSED AF Post-Approval Study
Status: Recruiting | Type: Observational
Sponsor: Medtronic Cardiac Ablation Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: PULSED AF PAS
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Paroxysmal: Ablation using the PulseSelect™ PFA system
  Interventions: Device: PulseSelect™ PFA system
- Persistent: Ablation using the PulseSelect™ PFA system
  Interventions: Device: PulseSelect™ PFA system

INTERVENTIONS:
Device: PulseSelect™ PFA system — Ablation using the PulseSelect™ PFA system

SUMMARY:
PULSED AF PAS is a prospective, global, multi-center, non-randomized, observational trial. Subjects will be treated with the PulseSelect™ PFA System and followed through 36 months.

DETAILED DESCRIPTION:
PulseSelect is a prospective, global, multi-center, non-randomized, observational trial. Subjects will be treated with the PulseSelect™ PFA System and followed through 36 months. Study visits will occur at 3, 6, 12, 24, and 36 months post-ablation, including required 24-hour Holter monitoring at 6, 12, 24, and 36 month visits. The PulseSelect™ PFA System used in this study is market approved and the ablation procedure will be performed according to hospital standard of care.

ELIGIBILITY:
Inclusion Criteria

* A diagnosis of recurrent symptomatic paroxysmal AF or persistent AF
* Refractory to at least one Class I or III antiarrhythmic drug (i.e., not effective, not tolerated, or not desired)
* Patient is ≥ 18 years of age
* Planned pulmonary vein isolation procedure with the commercially available PulseSelect™ PFA System
* Willing and able to comply with study requirements and give informed consent (defined as legally effective, documented confirmation of a subject's voluntary agreement to participate in this clinical study) or authorization per institution and geographical requirements

Exclusion Criteria

* Long-standing persistent AF (continuous AF sustained >12 months)
* Prior left atrial catheter or surgical ablation
* Patient with life expectancy < 36 months
* Presence of a permanent pacemaker, biventricular pacemaker, loop recorder/insertable cardiac monitor (ICM), or any type of implantable cardiac defibrillator (with or without biventricular pacing function)
* Current or anticipated participation in any other clinical trial of a drug, device, or biologic not approved by the global study manager

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects 18 years or older with a planned procedure using commercially available PulseSelect™ PFA System
Sampling Method: Non-Probability Sample
Enrollment: 580 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy-Freedom from Atrial Fibrillation | 36-months after the index ablation procedure
  Estimate the 36-month freedom from AF/AFL/AT recurrence following ablation using the PulseSelect™ PFA system.
Safety- Freedom from Device/Procedure Related Adverse Events | 6 months post-ablation]
  Estimate the rate of major procedural complications for catheter ablation using PulseSelect™ PFA system.

CONTACTS AND LOCATIONS:
Overall Officials: Khaldoun Tarakji, MD, Study Director — Medtronic CAS Chief Medical Officer
Locations (16):
- United States (16):
  - University of South Florida Health (USF), Tampa, Florida
  - Pikeville Medical Center, Whitesburg, Kentucky
  - Southcoast Health System, Fall River, Massachusetts
  - Beaumont Health System, Royal Oak, Michigan
  - Nebraska Medical Center, Omaha, Nebraska
  - The Valley Hospital, New York, New York
  - Northwell Health Lenox Hill Hospital, New York, New York
  - Duke University Medical Center (DUMC), Durham, North Carolina
  - Bethesda North Hospital, Cincinnati, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Mount Carmel Grove City Medical Center, Grove City, Ohio
  - Doylestown Health Cardiology a division of Doylestown Health Physicians, Doylestown, Pennsylvania
  - AnMed Health Center, Anderson, South Carolina
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Texas Health Research & Education Institute, Dallas, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia